CLINICAL TRIAL: NCT03971539
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses and Multiple Rising Oral Doses of BI 894416 Versus Placebo in Male Patients With Asthma (Single-blind, Randomised, Placebo-controlled, Parallel Group Design).
Brief Title: Evaluation of Safety and Tolerability of BI 894416 in Patients With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1371-0008; 2019-000805-60 (EudraCT Number)
Record Dates: First submitted 2019-05-20; First posted 2019-06-03 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- SRD part: Placebo (Placebo Comparator): Single rising dose (SRD) part: Placebo film-coated tablet matching BI 894416 taken once orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: Placebo
- SRD part: 75 mg BI 894416 (Experimental): Single rising dose (SRD) part: 75 milligram (mg) BI 894416 film-coated tablet taken once orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 894416; Drug: Placebo
- SRD part: 125 mg BI 894416 (Experimental): Single rising dose (SRD) part: 125 milligram (mg) BI 894416 film-coated tablet taken once orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 894416
- SRD part: 170 mg BI 894416 (Experimental): Single rising dose (SRD) part: 170 milligram (mg) BI 894416 film-coated tablet taken once orally with 240 milliliter of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 894416
- MRD part: Placebo (Placebo Comparator): Multiple rising dose (MRD) part: Placebo film-coated tablet matching BI 894416 taken for 9 days orally with 240 milliliter of water. Administration of Placebo at Day 1 and Day 9 once daily in the morning (q.d.) and at Day 2 to Day 8 three times daily at an interval of 8 hours (t.i.d.). Morning dose to be taken after an overnight fast of at least 10 hours, afternoon dose to be taken after fasting for 2 hours.
  Interventions: Drug: Placebo
- MRD part: 10 mg BI 894416 (Experimental): Multiple rising dose (MRD) part: 10 milligram (mg) BI 894416 film-coated tablet taken for 9 days orally with 240 milliliter of water. Administration of BI 894416 at Day 1 and Day 9 once daily in the morning (q.d.) and at Day 2 to Day 8 three times daily at an interval of 8 hours (t.i.d.). Morning dose to be taken after an overnight fast of at least 10 hours, afternoon dose to be taken after fasting for 2 hours.
  Interventions: Drug: BI 894416
- MRD part: 25 mg BI 894416 (Experimental): Multiple rising dose (MRD) part: 25 milligram (mg) BI 894416 film-coated tablet taken for 9 days orally with 240 milliliter of water. Administration of BI 894416 at Day 1 and Day 9 once daily in the morning (q.d.) and at Day 2 to Day 8 three times daily at an interval of 8 hours (t.i.d.). Morning dose to be taken after an overnight fast of at least 10 hours, afternoon dose to be taken after fasting for 2 hours.
  Interventions: Drug: BI 894416
- MRD part: 50 mg BI 894416 (Experimental): Multiple rising dose (MRD) part: 50 milligram (mg) BI 894416 film-coated tablet taken for 9 days orally with 240 milliliter of water. Administration of BI 894416 at Day 1 and Day 9 once daily in the morning (q.d.) and at Day 2 to Day 8 three times daily at an interval of 8 hours (t.i.d.). Morning dose to be taken after an overnight fast of at least 10 hours, afternoon dose to be taken after fasting for 2 hours.
  Interventions: Drug: BI 894416
- MRD part: 60 mg BI 894416 (Experimental): Multiple rising dose (MRD) part: 60 milligram (mg) BI 894416 film-coated tablet taken for 9 days orally with 240 milliliter of water. Administration of BI 894416 at Day 1 and Day 9 once daily in the morning (q.d.) and at Day 2 to Day 8 three times daily at an interval of 8 hours (t.i.d.). Morning dose to be taken after an overnight fast of at least 10 hours, afternoon dose to be taken after fasting for 2 hours.
  Interventions: Drug: BI 894416

INTERVENTIONS:
Drug: BI 894416 — BI 894416 film-coated tablet.
  Arms: MRD part: 10 mg BI 894416; MRD part: 25 mg BI 894416; MRD part: 50 mg BI 894416; MRD part: 60 mg BI 894416; SRD part: 125 mg BI 894416; SRD part: 170 mg BI 894416; SRD part: 75 mg BI 894416
Drug: Placebo — Placebo film-coated tablet matching BI 894416.
  Arms: MRD part: Placebo; SRD part: 75 mg BI 894416; SRD part: Placebo

SUMMARY:
In both parts, the primary comparisons of interest are between the percentage of patients with drug-related adverse events at each dose and placebo during single and multiple dosing regimens. Based on these, the primary trial objective is to assess safety and tolerability of BI 894416 at each dose.

Secondary measures of interest are the geometric means of BI 894416 plasma AUC0-∞ and Cmax after single dose in SRD part and AUC0-8 and Cmax after single dose as well as AUCτ,ss and Cmax,ss after 7 days multiple dosing in MRD part. The objective is to assess the pharmacokinetics of BI 894416 following single and multiple administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial. Medication washout and medication restrictions according to protocol are allowed only after informed consent is obtained.
* Male patients aged at least 18 years but not more than 55 years at the time of informed consent.
* Men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Pre-bronchodilator clinic measured FEV1 of ≥ 70% of predicted normal at the screening visit (Visit 1). Calculations will be based on Global Lung Function Initiative (GLI) formula
* A diagnosis of asthma, diagnosed by a physician.
* Patients should be non-smokers or ex-smokers who stopped smoking at least 12 weeks prior to screening and are expected to be able to not smoke for the duration of the study.
* Patients must be able to perform all trial related procedures including pulmonary function tests, nasal brushings.
* BMI of 18.5 to 32 kg/m2 (incl.)
* For MRD part: Patients are allowed to be on stable inhaled low dose corticosteroid (please refer to GINA guidelines) for at least 4 weeks prior to screening.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR, echocardiography and echocardiography stress test or ECG and including the neurological examination) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular (stress), metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug other than BI 894416 has been administered within 60 days or 5 half-lives (whichever is greater) prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug. In case of planned participation in the MRD part in this trial the previous participation in one dose group of the SRD part is allowed if BI 894416 has been administered more than 21 days prior to planned administration of BI 894416 in the MRD part. (Participation in an SRD dose group after the patient has participated in the MRD part is not allowed.)
* Alcohol abuse (consumption of more than 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Patient unable or unwilling to comply with study requirements, or has a condition that would not allow safe participation in the study
* History of relevant neurological disorder affecting the peripheral or central nervous system (this includes, but is not limited to: stroke, epilepsy, inflammatory or atrophic diseases affecting the nervous system, cluster headache or any cancer of the nervous system)
* History of immunological disease except allergy not relevant to the trial (such as mild hayfever or dust mite allergy) and except asthma in childhood or adolescence
* History of cancer (other than successfully treated basal cell carcinoma)
* Use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g. acetylsalicylic acid) within 10 days prior to administration of trial medication, or planned use during the trial or within 7 days after last dose of trial medication.
* Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer ITEM, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was randomised, placebo-controlled within groups, and single blinded. The trial consisted of a single rising dose (SRD) and a multiple rising dose (MRD) part. Last follow-up visit occurred between 14 and 16 days after the single dose for the SRD part and between day 14 and 21 days after the last dose for the MRD part.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | SRD Part: Placebo | SRD Part: 75 mg BI 894416 | SRD Part: 125 mg BI 894416 | SRD Part: 170 mg BI 894416 | MRD Part: Placebo | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416
Started | 6 | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Completed | 6 | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): the TS includes all patients who were randomised and treated with at least one dose of trial medication. The treatment assignment was determined based on the 1st treatment the patient received.
Groups:
- Total: Total of all reporting groups
Arm/Group | SRD Part: Placebo | SRD Part: 75 mg BI 894416 | SRD Part: 125 mg BI 894416 | SRD Part: 170 mg BI 894416 | MRD Part: Placebo | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416 | Total
Number analyzed (Participants) | 6 | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (12.3) | 30.6 (7.2) | 27.1 (7.5) | 29.3 (9.3) | 26.1 (4.4) | 32.7 (11.2) | 29.9 (10.6) | 30.9 (9.0) | 28.9 (9.0) | 30.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 7 | 8 | 7 | 8 | 7 | 7 | 8 | 8 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 5 | 7 | 8 | 8 | 8 | 7 | 7 | 8 | 7 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Treatment-emergent Adverse Events Related to BI 894416
Description: Percentage of patients with treatment-emergent adverse events (AEs) related to BI 894416.
Time Frame: From start of treatment till the end of trial, up to 30 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Groups:
- SRD Part: Total BI 894416: Single rising dose (SRD) part, total of all subjects treated with BI 894416 (75 mg, 125 mg and 170 mg).
- SRD Part: Total (BI 894416 and Placebo): Single rising dose (SRD) part, total of all subjects in SRD part (75 mg, 125 mg 170 mg and placebo).
- MRD Part: Total BI 894416: Multiple rising dose (MRD) part, total of all subjects treated with BI 894416 (10 mg, 25 mg, 50 mg and 60 mg).
- MRD Part: Total (BI 894416 and Placebo): Multiple rising dose (MRD) part, total of all subjects in MRD part (10 mg, 25 mg, 50 mg, 60 mg and placebo).
Arm/Group | SRD Part: Placebo | SRD Part: 75 mg BI 894416 | SRD Part: 125 mg BI 894416 | SRD Part: 170 mg BI 894416 | MRD Part: Placebo | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416 | SRD Part: Total BI 894416 | SRD Part: Total (BI 894416 and Placebo) | MRD Part: Total BI 894416 | MRD Part: Total (BI 894416 and Placebo)
Number analyzed (Participants) | 6 | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 23 | 29 | 31 | 39
Percentage of participants | 0 | 28.6 | 37.5 | 62.5 | 0.0 | 28.6 | 0.0 | 25.0 | 25.0 | 43.5 | 34.5 | 19.4 | 15.4

2. Secondary Outcome: AUC0-∞ (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity) of BI 894416 (SRD Part)
Description: AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) of BI 894416 (single rising dose part).
Time Frame: 3 hours before and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72 and 96 hours following treatment.
Population: Pharmacokinetic set (PKS): the PKS includes all patients in the TS who provided at least one pharmacokinetic endpoint that was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetics, or due to pharmacokinetic non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles*hours/liter
Arm/Group | SRD Part: 75 mg BI 894416 | SRD Part: 125 mg BI 894416 | SRD Part: 170 mg BI 894416
Number analyzed (Participants) | 7 | 8 | 8
Nanomoles*hours/liter | 15900 (41.5) | 26400 (30.0) | 32500 (21.9)

3. Secondary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma) of BI 894416 (SRD Part)
Description: Cmax (maximum measured concentration of the analyte in plasma) of BI 894416 (single rising dose part).
Time Frame: 3 hours before and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72 and 96 hours following treatment.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles/liter
Arm/Group | SRD Part: 75 mg BI 894416 | SRD Part: 125 mg BI 894416 | SRD Part: 170 mg BI 894416
Number analyzed (Participants) | 7 | 8 | 8
Nanomoles/liter | 2340 (29.7) | 4240 (25.3) | 5280 (24.3)

4. Secondary Outcome: AUC0-8 (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to 8 Hours) of BI 894416 After the First Dose (MRD Part)
Description: AUC0-8 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 8 hours) of BI 894416 after the first dose (Multiple rising dose part).
Time Frame: 5 minutes before and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6 and 8 hours following first dose (day 1).
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles*hours/liter
Arm/Group | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416
Number analyzed (Participants) | 7 | 8 | 8 | 8
Nanomoles*hours/liter | 992 (28.1) | 3130 (9.62) | 4320 (28.4) | 7310 (35.1)

5. Secondary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma) of BI 894416 After the First Dose (MRD Part)
Description: Cmax (maximum measured concentration of the analyte in plasma) of BI 894416 after the first dose (Multiple rising dose part).
Time Frame: 5 minutes before and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 23.92 hours following first dose (day 1).
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles/liter
Arm/Group | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416
Number analyzed (Participants) | 7 | 8 | 8 | 8
Nanomoles/liter | 239 (31.6) | 704 (20.6) | 1170 (40.0) | 1730 (49.5)

6. Secondary Outcome: AUCtau,ss (Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State) of BI 894416 After the Last Dose (MRD Part)
Description: AUCtau,ss (area under the concentration-time curve of the analyte in plasma at steady state) of BI 894416 after the last dose (Multiple rising dose part).
Time Frame: 5 minutes before and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours following last dose (day 9).
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles*hours/liter
Arm/Group | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416
Number analyzed (Participants) | 7 | 8 | 8 | 8
Nanomoles*hours/liter | 1460 (48.6) | 4770 (19.7) | 5420 (33.2) | 9400 (30.6)

7. Secondary Outcome: Cmax,ss (Maximum Measured Concentration of the Analyte in Plasma at Steady State) of BI 894416 After the Last Dose (MRD Part)
Description: Cmax,ss (maximum measured concentration of the analyte in plasma at steady state) of BI 894416 after the last dose (Multiple rising dose part).
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles/liter
Arm/Group | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416
Number analyzed (Participants) | 7 | 8 | 8 | 8
Nanomoles/liter | 299 (42.7) | 985 (19.4) | 1290 (52.1) | 2130 (30.3)

8. Secondary Outcome: Difference From Baseline in Airway Resistance (RAW) After 7 Days of Treatment (MRD Part)
Description: Difference in airway resistance (RAW) from baseline (measured on day 1) to day 9, after 7 days (day 2-8) of t.i.d. (three times daily) treatment.
Time Frame: Up to 9 days.
Population: Treated set (TS): the TS includes all patients who were randomised and treated with at least one dose of trial medication. The treatment assignment was determined based on the 1st treatment the patient received. The TS was used for safety analyses.
Measure: Mean (Standard Deviation); unit: kilopascal/liter/second
Arm/Group | MRD Part: Placebo | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 8
kilopascal/liter/second | 0.052 (0.086) | 0.069 (0.026) | 0.041 (0.038) | 0.041 (0.066) | 0.000 (0.082)

ADVERSE EVENTS:
Time Frame: From start of treatment till the end of trial, up to 30 days.
Description: Treated set (TS): the TS includes all patients who were randomised and treated with at least one dose of trial medication. The treatment assignment was determined based on the 1st treatment the patient received.
Groups:
- Total BI 894416: All subjects treated with BI 894416 in either the single rising dose or multiple rising dose part.
- Total: All subjects in the study.
Arm/Group | SRD Part: Placebo | SRD Part: 75 mg BI 894416 | SRD Part: 125 mg BI 894416 | SRD Part: 170 mg BI 894416 | MRD Part: Placebo | MRD Part: 10 mg BI 894416 | MRD Part: 25 mg BI 894416 | MRD Part: 50 mg BI 894416 | MRD Part: 60 mg BI 894416 | SRD Part: Total BI 894416 | SRD Part: Total (BI 894416 and Placebo) | MRD Part: Total BI 894416 | MRD Part: Total (BI 894416 and Placebo) | Total BI 894416 | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/8 | 0/8 | 0/8 | 0/7 | 0/8 | 0/8 | 0/8 | 0/23 | 0/29 | 0/31 | 0/39 | 0/54 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/8 | 0/8 | 0/8 | 0/7 | 0/8 | 0/8 | 0/8 | 0/23 | 0/29 | 0/31 | 0/39 | 0/54 | 0/68
Other Adverse Events (participants affected / at risk) | 1/6 | 5/7 | 5/8 | 7/8 | 6/8 | 5/7 | 7/8 | 7/8 | 5/8 | 17/23 | 18/29 | 24/31 | 30/39 | 41/54 | 48/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SRD Part: Placebo (N=6) | SRD Part: 75 mg BI 894416 (N=7) | SRD Part: 125 mg BI 894416 (N=8) | SRD Part: 170 mg BI 894416 (N=8) | MRD Part: Placebo (N=8) | MRD Part: 10 mg BI 894416 (N=7) | MRD Part: 25 mg BI 894416 (N=8) | MRD Part: 50 mg BI 894416 (N=8) | MRD Part: 60 mg BI 894416 (N=8) | SRD Part: Total BI 894416 (N=23) | SRD Part: Total (BI 894416 and Placebo) (N=29) | MRD Part: Total BI 894416 (N=31) | MRD Part: Total (BI 894416 and Placebo) (N=39) | Total BI 894416 (N=54) | Total (N=68)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 3 | 3
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Medical device site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Sluggishness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Mite allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Eyelid infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 2 | 4 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 2
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 3 | 4 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 4 | 7 | 3 | 1 | 0 | 3 | 3 | 13 | 13 | 7 | 10 | 20 | 23
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 2
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The planned last two dose level in the single rising dose (SRD) part and the last dose in the multiple rising dose (MRD) part were not used as the predicted exposure exceeded the limits predefined in the clinical trial protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03971539/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT03971539/SAP_001.pdf